CLINICAL TRIAL: NCT04075747
Title: V-FAST: A Phase 1b Master Trial to Investigate CPX-351 Combined With Various Targeted Agents in Subjects With Previously Untreated Acute Myeloid Leukemia
Brief Title: A Phase 1b Master Trial to Investigate CPX-351 in Subjects With Previously Untreated Acute Myeloid Leukemia
Acronym: V-FAST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZP025-101
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; venetoclax; midostaurin; enasidenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental)
  Interventions: Drug: CPX-351; Drug: Venetoclax
- Arm B (Experimental)
  Interventions: Drug: CPX-351; Drug: Midostaurin
- Arm C (Experimental)
  Interventions: Drug: CPX-351; Drug: Enasidenib

INTERVENTIONS:
Drug: CPX-351 — Up to 2 induction and 2 consolidation courses will be offered
  Other Names: Vyxeos; JZP351
Drug: Venetoclax — Will be administered over specified duration during induction and consolidation courses
  Other Names: Venclexta
  Arms: Arm A
Drug: Midostaurin — Will be administered over specified duration during induction and consolidation courses
  Other Names: Rydapt
  Arms: Arm B
Drug: Enasidenib — Will be administered over specified duration during induction and consolidation courses
  Other Names: Idhifa
  Arms: Arm C

SUMMARY:
JZP025-101 is an open-label, multicenter, multi-arm, nonrandomized phase 1b master trial to determine the recommended phase 2 dose (RP2D) of CPX-351 when administered in combination with various targeted agents in previously untreated subjects with Acute Myeloid Leukemia (AML) who are fit to receive intensive chemotherapy (ICT). Subjects will be assigned to treatment arms based on results of AML mutation testing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 to ≤ 75 years at the time of informed consent.
* Newly diagnosed AML according to World Health Organization (WHO) pathological criteria (with at least 20% blasts in the peripheral blood or bone marrow).
* ECOG performance status of 0 to 2.
* Laboratory values fulfilling the following:

  * Serum creatinine < 2.0 mg/dL.
  * Serum total bilirubin < 2.0 mg/dL. (For subjects with Gilbert's Syndrome and serum total bilirubin ≥ 2.0 mg/dL, the medical monitor should be contacted.)
  * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 times the upper limit of normal (ULN). (Note: If elevated liver enzymes > ULN are related to disease, contact medical monitor to discuss.)
* Cardiac ejection fraction ≥ 50% by echocardiography or multiple gated acquisition scan (MUGA).
* Subjects with second malignancies in remission may be eligible if there is clinical evidence of disease stability for a period > 6 months off cytotoxic chemotherapy, documented by imaging, tumor marker studies, etc., at screening. Subjects maintained on long-term nonchemotherapy treatment (eg, hormonal therapy) are eligible.

Exclusion Criteria:

* Acute promyelocytic leukemia [t(15;17)].
* Subject has favorable risk cytogenetics ((t8;21), inv(16), t(16;16), or t15;17) karyotype abnormalities) as categorized by the National Comprehensive Cancer Network (NCCN) Guidelines Version 2.2014 for AML (NCCN 2014).
* Clinical evidence of active central nervous system (CNS) leukemia.
* Subjects with active (uncontrolled, metastatic) second malignancies.
* Subjects who have received prior treatment intended for induction therapy of AML; only hydroxyurea is permitted for control of blood cell counts. (For example, a subject with myelodysplastic syndrome [MDS] who changes hypomethylating agent [HMA] dose and schedule after the diagnosis of AML is excluded. AML-type therapy, such as cytarabine alone [> 1g/m2/day] or cytarabine plus an anthracycline as well as prior HSCT are also excluded.) All-trans-retinoic acid (ATRA) used empirically is permitted.
* Subjects receiving administration of any therapy for MDS (conventional or investigational) must be completed by 2 weeks prior to the first dose of study drug. In the event of rapidly proliferative disease, use of hydroxyurea is permitted until 24 hours before the start of study treatment. Toxicities associated with prior MDS therapy must have recovered to Grade 1 or less prior to start of treatment.
* Subjects with myocardial impairment of any cause (eg, cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging).
* Subjects with active or uncontrolled infection. Subjects with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥ 72 hours.
* Current evidence of invasive fungal infection (blood or tissue culture). Subjects with recent fungal infection must have a subsequent negative culture to be eligible.
* Subjects with known human immunodeficiency virus (new testing not required) or evidence of active hepatitis B or C infection.
* Subjects with known history of Wilson's disease or other known copper-metabolism disorder.
* Subjects with other comorbidity that the investigator judges to be incompatible with conventional ICT, and / or the targeted agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Determine the Recommended Phase 2 Dose (RP2D) | Up to 30 months
  The RP2D will be determined by the specified dose de-escalation/dose escalation algorithm.
Safety and Tolerability of CPX-351 and Targeted Agents: incidence of adverse events (AEs) and dose limiting toxicities (DLTs) | Up to 30 months
  The safety and tolerability of CPX-351 and targeted agents when given in combination, based on the incidence of adverse events (AEs) and dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Proportion of subjects who have achieved CR, CRi, CRh, CR + CRi, CR + CRh, and morphologic leukemia-free state (MLFS) | Up to 30 months
  After up to 2 inductions
Proportion of subjects who have achieved CR / CRi with MRD negative status | Up to 30 months
  After up to 2 inductions
Proportion of subjects who have achieved CR / CRh with MRD negative status | Up to 30 months
  After up to 2 inductions

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - Stanford University School of Medicine- Standford Cancer Institute, Palo Alto, California
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University of Kansas Cancer Center, Fairway, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University, Durham, North Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pullarkat VA, Levis M, McCloskey J, Mannis GN, Strickland SA, Fathi AT, Lin TL, Bhatt VR, Vanniyasingam T, Chakravarthy D, Lutska Y, Faderl S, Cheung RS, Erba HP. V-FAST: a phase 1b master trial to investigate CPX-351 combined with targeted agents in adults with newly diagnosed AML. Blood Neoplasia. 2025 Jun 3;2(4):100123. doi: 10.1016/j.bneo.2025.100123. eCollection 2025 Nov. PMID 40932876